CLINICAL TRIAL: NCT00049530
Title: Phase II Study of Low Dose Peginterferon Alfa-2b in Patients With Metastatic Melanoma Over-Expressing Basic Fibroblast Growth Factor
Brief Title: PEG-Interferon Alfa-2b in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258114; E2602 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-interferon alfa-2b (Experimental): Patients receive PEG-interferon alfa-2b subcutaneously (SC) once weekly. Treatment continues until basic fibroblast growth factor level is suppressed to normal or until a maximum weekly dose is reached. If there is disease progression, patients then discontinue treatment. If there is no disease progression, patients receive PEG-interferon alfa-2b SC weekly for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: PEG-interferon alfa-2b

INTERVENTIONS:
Biological: PEG-interferon alfa-2b — Patients receive PEG-interferon alfa-2b subcutaneously (SC) once weekly. Treatment continues until basic fibroblast growth factor level is suppressed to normal or until a maximum weekly dose is reached. If there is disease progression, patients then discontinue treatment. If there is no disease progression, patients receive PEG-interferon alfa-2b SC weekly for up to 1 year in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Peginterferon (PEG-interferon) alfa-2b may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of PEG-interferon alfa-2b in treating patients who have stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of low-dose PEG-interferon alfa-2b to suppress plasma basic fibroblast growth factor (b-FGF) levels to normal in patients with metastatic melanoma over-expressing b-FGF.
* Determine the antitumor effect of this drug, in terms of progression-free and overall survival and tumor response, in these patients.
* Correlate tumor activity of this drug with b-FGF and vascular endothelial growth factor levels in the plasma and urine of these patients.
* Determine the safety profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive PEG-interferon alfa-2b subcutaneously (SC) once weekly. Treatment continues until basic fibroblast growth factor level is suppressed to normal or until a maximum weekly dose is reached. If there is disease progression, patients then discontinue treatment. If there is no disease progression, patients receive PEG-interferon alfa-2b SC weekly for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion criteria:

* Histologically confirmed stage IV melanoma

  * Stage M1a, M1b, or M1c
  * Mucosal, ocular, or unknown primary melanoma
* Previously untreated OR received up to 3 prior systemic therapy regimens (excluding vaccine therapy) for metastatic disease
* Plasma basic fibroblast growth factor level at least 15 pg/mL
* Measurable or evaluable disease
* Central nervous system (CNS) involvement allowed provided CNS directed therapy has been given and disease has been clinically stable for ≥ 3 months

  * Brain computed tomography (CT) scan or Magnetic resonance imaging (MRI) to confirm stable disease required ≤ 4 weeks prior to study entry
* Age: 18 and over
* ECOG Performance status of 0-2
* Life expectancy at least 6 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL (transfusions allowed)
* Bilirubin no greater than 2 times upper limit of normal (ULN)
* Alanine Aminotransferase (ALT) no greater than 2 times ULN
* Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min
* At least 4 weeks since prior interferon in the adjuvant or metastatic setting
* At least 4 weeks since prior chemotherapy in the adjuvant or metastatic setting
* At least 4 weeks since prior endocrine therapy in the adjuvant or metastatic setting
* At least 4 weeks since prior radiotherapy in the adjuvant or metastatic setting
* At least 4 weeks since prior surgery in the adjuvant or metastatic setting
* At least 4 weeks since other prior therapy in the adjuvant or metastatic setting
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Myocardial infarction within the past 6 months
* Other active malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* Other concurrent illness that would preclude study participation
* History of severe depression
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-01-13 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S. Go, MD, Study Chair — Gundersen Lutheran Center for Cancer and Blood
Locations (32):
- United States (32):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on September 5, 2003, accrued its first patient on January 13, 2004, and patient accrual was terminated on June 15, 2011. A total of 32 patients were enrolled through ECOG member institutions. The study was suspended three times during the accrual period (February 2005, November 2006, January 2009) due to unavailability of ELISA kits to measure fibroblast growth factor.
Pre-assignment Details: This study involves a pre-registration and a registration. In the pre-registration phase, plasma samples must be submitted for determinations of b-FGF status by central analysis. Only patients determined to have an elevated b-FGF level (>15 pg/mL) by central review are eligible for registration.
Period: Overall Study
Arm/Group | PEG-interferon Alfa-2b
Started | 32
Eligible and Treated | 29
Completed | 0
Not Completed | 32
Not completed — Lack of Efficacy | 25
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — symptomatic deterioration | 1
Not completed — ineligible | 3

BASELINE CHARACTERISTICS:
Population: The primary analysis population was all eligible (meeting all eligibility criteria listed in protocol) and treated patients (receiving at least one dose of the protocol therapy). All baseline analysis and efficacy endpoints are based on the primary population (n=29).
Arm/Group | PEG-Interferon Alfa-2b
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 64 [39 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Plasma b-FGF Level Response
Description: The primary endpoint was the suppression of plasma b-FGF level with low dose peginterferon alfa-2b. A clinically important reduction of plasma b-FGF levels was determined to be a level less than or equal to 7.5 pg/mL. A patient was considered to have a suppressed plasma b-FGF level, if the patient experienced the clinically significant reduction (less than or equal to 7.5 pg/mL) of plasma b-FGF levels for two consecutive determinations which were at least three weeks apart. This was considered as a b-FGF response.
Time Frame: assessed every 3 weeks until the suppression of plasma b-FGF level to normal, then every 6 weeks until the completion of 12 months of treatment, and upon treatment discontinuation
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-interferon Alfa-2b
Number analyzed (Participants) | 29
percentage of participants | 34.5 [17.9 to 54.3]
Statistical Analysis 1: Comparison: PEG-interferon Alfa-2b; It is of interest to test the null hypothesis of 10% plasma b-FGF response rate versus the alternative hypothesis of 30% response rate. Based on the sample size of 30 eligible patients, there will be 84% power to detect this 20% difference in b-FGF response rates. This was based on a two-sided type I error of .05, using the one-sample binomial test; Test type: Superiority or Other; p < 0.001, bionomial proportion test

2. Secondary Outcome: Non-progression Rate (Clinical Response to Peginterferon Alfa-2b)
Description: Objective tumor response was assessed using RECIST (Response Evaluation Criteria in Solid Tumors) 1.0 criteria. Per RECIST criteria, complete response (CR) = disappearance of all target and non-target lesions. Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits. Progression is defined as at least 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum longest diameter recorded since the baseline measurements, or the appearance of one or more new lesion(s) or unequivocal progression of existing non-target lesions. Stable disease (SD) = did not meet criteria for response or progression.
  Non-progression rate = CR + PR + SD.
Time Frame: assessed every 9 weeks until suppression of plasma b-FGF level to normal, every 12 weeks until the completion of 12 months of treatment, >= 4 weeks after documented response. After off treatment, every 3 months if <2 years, and every 6 months if 2-3 years
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PEG-interferon Alfa-2b
Number analyzed (Participants) | 29
percentage of participants | 24.1 [10.3 to 43.5]

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the time from registration to disease progression, or censored at last known date of non progressive disease.
Time Frame: as for outcome 2
Population: eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PEG-interferon Alfa-2b
Number analyzed (Participants) | 29
months | 2 [1.8 to 2.3]

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) time was defined as the time from registration to death from any cause, or censored at last known date of survival.
Time Frame: assessed every 3 months if <2 years, and every 6 months if 2-3 years
Population: eligible and treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PEG-interferon Alfa-2b
Number analyzed (Participants) | 29
months | 9.7 [4.4 to 12.5]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks in induction phase, every 6 weeks in maintenance phase, and for 30 days after the end of treatment, up to 3 years.
Description: Adverse events occurred within 30 days after the end of treatment were reported in the Adverse Event Form for the last cycle. Long term grade 3 or higher adverse event which has not been previously reported were also included in the reporting (assessed every 3 months if patient is <2 years from study entry and every 6 months if 2-3 years).
Arm/Group | PEG-Interferon Alfa-2b
Serious Adverse Events (participants affected / at risk) | 13/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-Interferon Alfa-2b (N=32)
Anemia (Blood and lymphatic system disorders) | 1
White blood cell decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Hypotension (Vascular disorders) | 1
Fatigue (General disorders) | 7
Chills (General disorders) | 1
General disorders and administration sit (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 1 — details were unknown (no data)
Alanine aminotransferase increased (Investigations) | 1
Infections w/o neutropenia (Infections and infestations) | 2
Confusion (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Tremor (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-Interferon Alfa-2b (N=32)
Anemia (Blood and lymphatic system disorders) | 15
White blood cell decreased (Investigations) | 12
Neutrophil count decreased (Investigations) | 12
Platelet count decreased (Investigations) | 6
Fatigue (General disorders) | 24
Fever (General disorders) | 11
Chills (General disorders) | 6
Weight loss (Investigations) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Injection site reaction (General disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 15
Constipation (Gastrointestinal disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 13
Dysgeusia (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 4
Blood bilirubin increased (Investigations) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alanine aminotransferase increased (Investigations) | 10
Dizziness (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 4
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 5
Nervous system disorders - Other, specif (Nervous system disorders) | 2 — details were unknown (no data)
Tremor (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 4
General disorders and administration sit (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No